CLINICAL TRIAL: NCT06510348
Title: Achieving nuTritional Target in criticAlly Ill patieNts With iMpairEd gastroiNtesTinal Dysfunction
Acronym: ATTAINMENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Romanian Society for Enteral and Parenteral Nutrition (Other)
Collaborators: Fresenius Kabi (Industry); Carol Davila University of Medicine and Pharmacy (Other); Bucharest Emergency Hospital (Other)
Responsible Party: Principal Investigator, Cristian Cobilinschi, Principal Investigator, MD, PhD,, Romanian Society for Enteral and Parenteral Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATTAINMENTstudy
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Parenteral Nutrition; Gastroparesis; Gastrointestinal Dysfunction; Protein Deficiency; Critical Illness
Keywords: gastrointestinal dysfunction; supplemental parenteral nutrition; parenteral nutrition; enteral nutrition; critically ill; protein intake; calorie intake; gastroparesis; malabsorption
MeSH Terms: conditions — Hyperphagia; Gastroparesis; Protein Deficiency; Critical Illness; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EN group (No Intervention): enteral nutrition intake will progressively be increased according to the gastrointestinal tolerance (evaluated based on ultrasound guided gastric residual volume measurement) until the target of 100% is attained following admission to the ICU.
- Supplemental parenteral nutrition (SPN) group (Experimental): gradually initiate supplemental parenteral nutrition in order to achieve the target of 80% by the fifth day. Trophic feed will be administered to cover the remaining 20% of the targeted nutrition intake.
  Interventions: Dietary Supplement: Supplemental Parenteral Nutrition (SPN)

INTERVENTIONS:
Dietary Supplement: Supplemental Parenteral Nutrition (SPN) — Nutritional targets are based on ESPEN guidelines recommendation (calories administration based on indirect calorimetry study, proteins 1.3 g/kg/day). From the first day of ICU admission indirect calorimetry will be performed daily in order to evaluate energy requirements. On the fourth day, the patient will undergo a gastric residual volume measurement and a paracetamol absorption test. If gastrointestinal dysfunction is detected, the patient will be assigned to a study group based on the randomization protocol. The SPN group will gradually initiate supplemental parenteral nutrition in order to achieve the target of 80% by the fifth day. Trophic feed will be administered to cover the remaining 20% of the targeted nutrition intake.
  Arms: Supplemental parenteral nutrition (SPN) group

SUMMARY:
Clear study hypothesis / research question

It has already been proven that a prolonged negative energy balance during intensive care stay is an independent risk factor for mortality. Although it was thought that achivieng optimal delivery of calories will prevent nutritional deficits in critically ill patients, published randomized controlled trials failed to confirm this hypothesis.

Combinging enteral and parenteral support may be an efficent strategy to reach nutritional target in critically ill patients. According to the current guidelines the use of suplemental parenteral nutrition (SPN) should be considered when energy targets are not achieved by enteral (EN) route, however, no clear data regarding timing, amount and composition is specified. Moreover, based on recente published data overfeeding should also be avoided, considering the negative impact on outcome.

Nutritional support for critically ill patients was focused more on preventing caloric and protein deficits and no great emphasis was placed on the efficiency of intestinal absorption. Gastrointestinal dysfunction is a prevalent reported complication that may contribute to falling short of meeting nutritional goals. This encompasses a wide spectrum of symptoms, such as impaired gastric emptying, ileus or impaired intestinal absorbtion, exposing patients to feeding intolerance, malnutrition and worse outcomes. No standard definition and monitoring techniques are so far available for the diagnostic of feeding intolerance. Although increased gastric residual volume (GRV) is the most used parameter for highlighting feeding intolerance, a controversy regarding the adequate threshold of GRV persists. Acetaminophen absorption test has been previously proposed as a diagnostic tool to asses impaired gastric emptying and intestinal absorbtion.

Besides intestinal absorbtion, efficient utilization of macronutients should also be assessed, considering that critically ill patients have varying metabolic conditions and may not be able to metabolically handle adminsitered substrates. As a result body composition analysis should be taken into account in order to obtain a dynamic quantification, especially, of the mucle mass compartiments.

Therefore the following low-interventional study is designed to investigate the hypothesis regarding energy and protein intake achievement in critically ill patients with diagnosed impaired gastrointestinal dysfunction to whom tailored nutritional support is administered.

Taking into account that we aim to identify patients with early-phase gastrointestinal dysfunction impaired gastric emptying and reduced intestinal absorbtion (diagnosed using ultrasound gastric residual volume and byacetaminiphen absorbtion test) will serve as defining factors. Patients will be randomized to receive nutritional support either according to the EN protocol or enteral trophic feed + SPN protocol.

Differences in rectus femoris thickness measured on admission, on day 10 and 15, variation of lean body mass measured by bioelectrical impedance on admission on day 10 and 15, and differences between groups in muscle function using handgrip dynamometer will also be evaluated in both groups.

DETAILED DESCRIPTION:
Rationale and clinical significance of the hypothesis

It has already been stated that nutritional support represents a crucial component in the care of critically ill patients. High metabolic demand encountered for critically ill patients may cause significant energy deficits responsible for increased risk of infection, prolonged mechanical ventilation and ICU stay. Aditionally, providing nutritional support in ICU patients is often deeemd challenging, as enteral feeding intolerance devolps secondary to gastrointestinal dysfunction. Although some authors opinioned that reducing energy targets might be beneficial, several studies proved that permissive underfeeding has no positive impact on outcome. Morover, reduction of energy target recommendation was associated with a scondary decrease of protein supplementation.

Apart from disscussing nutritional intake, great emphasis should be placed on nutritional uptake as an increased percentage of critically ill patients fail to reach nutritional targets often due to gastrointestinal dysfunction.

Gastrointestinal dyfunction may be defined by a variety of functional impairements affecting motility, absorbtion, microbiome composition or perfusion, but still, at this momement there is a lack of recommendation regarding monitoring methods[6]. At the bedside, assesement of gastrointestinal dysfunction often relies on measuring GRV. However, gastric emptying rate proved to be poorly correlated with GRV. This monitoring technique may also result in a decresed amount of nutrients delivery. Since ultrasound has became a popular diagnostic tool also in the ICU, several studies indicated that ultrasonographic measurement of gastric antral cross-sectional area has a good correlation with both aspirated GRV and gastric volume measured by computerised tomography. Considering that paracetamol has little to no absorption in the stomach and is completely absorbed at the intestinal level, paracetamol absorption test (PAT) has been proposed as a simple, indirect method for evaluating gastric emptying. As the pharmacokinetic studies have established that gastric emptying is a rate-limiting step for paracetamol absorbtion, studies where PAT was used, validated a significant correlation with scintigraphy results.

The combination of reduced tolerance to enteral feeding at the initiation of nutritional support, along with the initiation of nutritional support within 48 hours, has been proven to be responsible for a progressively significant and intractable energy deficit. It has been found that continuing enteral feeding under these circumstances is ineffective in resolving this energy debt which is proportional with an increased risk of nosocomial infections.

Using SPN for patients who cannot tolerate EN proved to be safe and was associated with improved cumulative energy balance, decreased rate of infections and significant cost reduction. Although SPN is proposed both by ESPEN and ASPEN guideline as an efficient alternative when energy and protein target are not achieve by oral or enteral route, recent data revealed that SPN use is rather limited[14]. The primary concern regarding SPN use is the risk of overfeeding. However, utilizing the appropriate concept of SPN and measuring energy needs by indirect calorimetry may overcome administering feeds in an unphysiological manner.

Besides intake and uptake, muscle capacity to respond to nutritional protein should also be taken into account. Several different tools have been proposed for body composition analysis of critically ill patients. Ultrasound with different protocols has also been used to assess muscle mass even in ICU patients with greater fluid shifts[16]. Studies have indicated that a significant reduction in muscle mass may be identified by both rectus femoris cross-sectional area and quadriceps muscle layer thickness measurements. Bioelectrical impedance analysis is another non-invasive, low-cost technique used for body composition assesment. Despite reported limitations related with frequent overhydration states in critically ill patients, this method can still provide reliable data if the appropriate timing for examination is chosen. Nevertheless, bioelectrical impedance analysis-derived phase angle proved to be a trustworthy parameter not only for evaluating fat-free mass, but also mortality. Functional parameters, such as handgrip strengts measurements should be also included when effectivness of nutritional support is evaluated. However, it is important to acknowledge barriers to collecting functional outcome data particularly when critically ill patients are studied.

Study design

1. Study type This single-center controlled randomized pragmatic trial will be conducted in the 34-bed general intensive care of Clinical Emergency Hospital of Bucharest, a tertiary-care university affiliated hospital.

   Participating site data:

   Department of Anaesthesia and Intensive Care from the Clinical Emergency Hospital of Bucharest disposes in total of 86 intensive care beds

   Considering that there is no globally validated single definition that can be used to objectify this gastrointestinal dysfunction, real prevalence of this dysfunction is not quantified. It has been reported that one-third of all enterally fed, mechanically ventilated, critically ill patients are presenting enteral feed intolerance, but many more patients may have subclinical gastrointestinal dysmotility, the estimated percentage could reach as high as 80%. Taking into account the annual rate of admission in our unit it is feasible to complete the inclusion process by July 2025 (1 year and 8 months).

   Nevertheless, maintaining this study as monocentric will provide better control over potential confounding factors and reduce heterogeneity. Furthermore, it will enhance internal validity and streamline coordination efforts.

   Ethics:

   Study protocol together with a a model of informed consent were submitted to the Clinical Emergency Hospital of Bucharest Ethics Committee and the final approval has been obtained on 18.05.2023.

   Taking into account that the included patients are not able to provide informed consent at the time of recruitment (on ICU admission), a Power of Attorney or a Legal tutor will act as Consultee and will be asked to consent/decline participation to the study on legal behalf of the patient. If patients have Advance Decision Plan including participation in research studies the Plan will be respected and recruitment pursued/abandoned accordingly. After regaining capacity, all patients will be asked to provide Informed Consent for using their personal data and will be given the possibility to:

   Provide Informed Consent for the acute data and follow-up. Deny research participation and request destruction of acute data collected.
2. Description of the study population (inclusion and exclusion criteria)

All adults (> 18 years old) are eligible for inclusion if it will be expected to require mechanical ventilation for more than four days, have a controlled shock state (hemodynamic and tissue perfusion goals are reached) and impaired intestinal absorbtion, defiend by both ultrasound measurement of gastric residual volume and paracetamol absorbtion test. Exclusion criteria are patients on non-invasive mechanichal ventilation, contraindication for EN for > 48 h after admission, patients with gastrointestinal surgical intervention within 3 months, history of malabsorption, inflammatory bowel disease, short bowel syndrom, anorexia nervosa, gastrointestinal bleeding, cirrhosis, traumatic brain injury, subarahnoidal hemorrhage, neoplasia, post cardiac arrest patients, patients on chronic therapy with corticosteroids and pregnant women.

e. Methods and techniques

Randomisation:

Selected patients for inclusion will be allocated in one of the two groups after stratified randomisation.

The patient population can be stratified into three groups based on their admission type, which includes General Surgery, Multiple Trauma, and Internal Medicine. To perform stratified randomization, three separate randomization lists would be required - one for each stratum. These lists could be generated using techniques such as block randomization. Depending on the stratum a patient belongs to, the corresponding randomization list would be utilized to allocate the patient to one of the nutritional protocol being compared.

Nutritional protocol:

Nutritional targets are based on ESPEN guidelines recommendation (calories administration based on indirect calorimetry study, proteins 1.3 g/kg/day). From the first day of ICU admission indirect calorimetry will be performed daily in order to evaluate energy requirements. For both groups enteral nutritional support will be started after 48 hours since admission or after controlled shock state will be confirmed. Enteral nutrition will be incrementally escalated using a ramped fashioned approach, with the goal of reaching 25 to 50% of the energy target determined by indirect calorimetry by day 2. Subsequently, on days 3 and 4, the target will be gradually raised to 75%. Enteral nutrition will be administered continuously.

On the fourth day, the patient will undergo a gastric residual volume measurement and a paracetamol absorption test. If gastrointestinal dysfunction is detected, the patient will be assigned to a study group based on the randomization protocol.

In the EN group, enteral nutrition intake will progressively be increased according to the gastrointestinal tolerance (evaluated based on ultrasound guided gastric residual volume measurement) until the target of 100% is attained following admission to the ICU.

The SPN group will gradually initiate supplemental parenteral nutrition in order to achieve the target of 80% by the fifth day. Trophic feed will be administered to cover the remaining 20% of the targeted nutrition intake. Figure 1 depicts a graphical illustration of the nutritional protocol.

Products:

EN formula for EN group and trophic feeds: polymeric, fibre-enriched formulas - Fresubin® Original Fibre (15% proteins, 30% lipids, 52% carbohydrates, Fibre 3 %) PN formula for SPN group: SMOFKABIVEN EXTRA NITROGEN 16 gN - 1518 ml - 10% amino acids, 20% lipid emulsion (SMOFlipid 20%), 42% glucose, and electrolytes

Ultrasound guided gastric residual volume measurement:

Gastric ultrasound assessment will be performed by two independent observers in supine position. Both sets of measurements will be performed after a minimum of six hours of fasting. Antral cross-sectional area (ACSA) area will be calculated by using antero-posterior and cranio-caudal antral diameters (measured from serosa to serosa) and the formula of the area of an elipse ( )/4). Furthermore, the gastric volume will be calculated according to the model proposed by Perlas et al. Gastric Volume (ml) = 27.63 + 0.16 x weight (kg) + 1.24 x BMI - 0.013 x (time since last meal in hours) x (antral cross-sectional area in cm²).

A gastric residual volume above 200 ml will be considered positive for impaired gastric motility.

Paracetamol absorbtion test:

In order to evaluate paracetamol absorbtion, area under the plasma concentration curve was chosen to be calculated at 240 mins (AUC240) by using the trapezoidal method. In order to be able to obtain AUC240 five different measurements will be carried out at predetermined intervals, namely at the baseline (before paracetamol administration), at 30 minutes, 60 minutes, 120 minutes, and 240 minutes. Paracetamol 15 mg/kg disolved in 10 ml aqueous solution followed by 20 ml of water will be adminsitered.

Afterwards Enzyme Multiplied Immunoassay Technique (EMIT) will be used to detect paracetamol level.

Principle of technique: The technique involves conjugating an enzyme with a small target molecule specific to the analyte being tested, in this case acetaminophen. Binding of a specific target antibody inhibits the enzymatic activity. The enzyme glucose-6-phosphate dehydrogenase is bound to the antigen for acetaminophen, which oxidizes glucose-6-phosphate to gluconolactone-6-phosphate and reduces NAD to NADH. If a free target molecule such as acetaminophen is present in the plasma, inhibition is weakened by competition for the antibody, leading to restoration of enzymatic activity and intensity of the signal proportional to the concentration of the free target molecule. Enzymatic activity is measured by spectroscopic analysis of the amount of NADH produced, which correlates directly to the amount of acetaminophen in the specimen. Blood samples will be collected from patients in vacutainer tubes with sodium citrate or EDTA anticoagulant under vacuum to facilitate plasma separation and prevent hemolysis.

Bioelectrical impedance analysis (BIA):

We will use the InBody BWA 2.0 BIA machine to perform BIA measurements. The following measurements will be collected for analysis: impedance, phase angle, resistance, reactance, Waist/Hip Ratio, body cellular mass, lean body mass and fat-free mass index.

Measurement of rectus femoris cross sectional area:

B-mode ultrasonography utilizing an 8 MHz 5.6 cm linear transducer array will be employed to measure the Cross-sectional area of the rectus femoris (RFCSA), employing a previously described technique. The transducer will be positioned perpendicularly to the long axis of the thigh, on its superior aspect, specifically three-fifths of the way from the anterior superior iliac spine to the superior patellar border.

ELIGIBILITY:
Inclusion Criteria:

* All adults (> 18 years old)
* Mechanical ventilation for more than four days,
* Controlled shock state (hemodynamic and tissue perfusion goals are reached) - Impaired intestinal absorbtion, defiend by both ultrasound measurement of gastric residual volume and paracetamol absorbtion test

Exclusion Criteria:

* patients on non-invasive mechanichal ventilation
* contraindication for EN for > 48 h after admission
* patients with gastrointestinal surgical intervention within 3 months,
* history of malabsorption, inflammatory bowel disease
* short bowel syndrom
* anorexia nervosa
* gastrointestinal bleeding
* cirrhosis
* traumatic brain injury
* subarahnoidal hemorrhage
* neoplasia
* post cardiac arrest patients
* patients on chronic therapy with corticosteroids
* pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the attainment (in percentage) of daily calorie | day 15
  Differences in the attainment (in percentage) of daily calorie pre-set targets* calculated from the rest energy expenditure measured (mREE) using indirect calorimetry (IC) between the EN and SPN groups.
  *pre-set targets are defined according to the described nutritional protocol (see below Section e. Nutritional protocol) as 25 % of the energy target determined by indirect calorimetry by day 2, 50% by day 3 to 4 and 75 % at day 4. After day 4 the pre-set target is gradually increased to 100 %.
Differences in the attainment (in percentage) of daily protein | day 15
  Differences in the attainment (in percentage) of daily protein pre-set targets* calculated from the rest energy expenditure measured (mREE) using indirect calorimetry (IC) between the EN and SPN groups.
  *pre-set targets are defined according to the described nutritional protocol (see below Section e. Nutritional protocol) as 25 % of the energy target determined by indirect calorimetry by day 2, 50% by day 3 to 4 and 75 % at day 4. After day 4 the pre-set target is gradually increased to 100 %.

SECONDARY OUTCOMES:
Differences in rectus femoris thickness measured on admission, on day 10 and 15 | day 15
  ultrasound measurement
Variation of phase angle between two groups | day 15
  measured by bioelectrical impedance analysis
Variation of lean body mass measured by bioelectrical | day 15
  measured by bioelectrical impedance analysis
muscle force measured on day 15 | day 15
  using handgrip dynamometer
energy adequacy | day 15
  Energy adequacy (%) = ratio between sum of percentage calories received/prescribed each day/ total number of evaluable nutrition days
protein adequacy | day 15
  Protein adequacy (%) = ratio between sum of percentage proteins received/prescribed each day/ total number of evaluable nutrition days
Mortality | on day 28
  dead or alive on day 28
ureea/creatinine ratio | on day 15
blood glucose concentration | on day 15
insulin rate | day 15

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Cobilinschi, MD, PhD, Principal Investigator — Bucharest Emergency Hospital; Liliana Mirea, Md PhD, Study Director — Bucharest Emergency Hospital; Radu Tincu, MD PhD, Study Chair — Bucharest Emergency Hospital; Ioana Grințescu, Profesor, Study Chair — Carol Davila University of Medicine and Pharmacy
Locations (1):
- Clinical Emergency Hospital of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger MM, Soguel L, Charriere M, Theriault B, Pralong F, Schaller MD. Impact of the reduction of the recommended energy target in the ICU on protein delivery and clinical outcomes. Clin Nutr. 2017 Feb;36(1):281-287. doi: 10.1016/j.clnu.2015.12.002. Epub 2015 Dec 28. PMID 26775753
- [Result] Chapman MJ, Deane AM. Gastrointestinal dysfunction relating to the provision of nutrition in the critically ill. Curr Opin Clin Nutr Metab Care. 2015 Mar;18(2):207-12. doi: 10.1097/MCO.0000000000000149. PMID 25603226
- [Result] Berger MM, Pantet O, Jacquelin-Ravel N, Charriere M, Schmidt S, Becce F, Audran R, Spertini F, Tappy L, Pichard C. Supplemental parenteral nutrition improves immunity with unchanged carbohydrate and protein metabolism in critically ill patients: The SPN2 randomized tracer study. Clin Nutr. 2019 Oct;38(5):2408-2416. doi: 10.1016/j.clnu.2018.10.023. Epub 2018 Nov 5. PMID 30448193
- [Result] Berger MM, Burgos R, Casaer MP, De Robertis E, Delgado JCL, Fraipont V, Goncalves-Pereira J, Pichard C, Stoppe C. Clinical nutrition issues in 2022: What is missing to trust supplemental parenteral nutrition (SPN) in ICU patients? Crit Care. 2022 Sep 10;26(1):271. doi: 10.1186/s13054-022-04157-z. PMID 36088342
- [Result] Toledo DO, Freitas BJ, Dib R, Pfeilsticker FJDA, Santos DMD, Gomes BC, Silva-Jr JM. Peripheral muscular ultrasound as outcome assessment tool in critically ill patients on mechanical ventilation: An observational cohort study. Clin Nutr ESPEN. 2021 Jun;43:408-414. doi: 10.1016/j.clnesp.2021.03.015. Epub 2021 Apr 6. PMID 34024548
- [Result] Moonen HPFX, Van Zanten ARH. Bioelectric impedance analysis for body composition measurement and other potential clinical applications in critical illness. Curr Opin Crit Care. 2021 Aug 1;27(4):344-353. doi: 10.1097/MCC.0000000000000840. PMID 33967207
- [Result] Reintam Blaser A, Preiser JC, Fruhwald S, Wilmer A, Wernerman J, Benstoem C, Casaer MP, Starkopf J, van Zanten A, Rooyackers O, Jakob SM, Loudet CI, Bear DE, Elke G, Kott M, Lautenschlager I, Schaper J, Gunst J, Stoppe C, Nobile L, Fuhrmann V, Berger MM, Oudemans-van Straaten HM, Arabi YM, Deane AM; Working Group on Gastrointestinal Function within the Section of Metabolism, Endocrinology and Nutrition (MEN Section) of ESICM. Gastrointestinal dysfunction in the critically ill: a systematic scoping review and research agenda proposed by the Section of Metabolism, Endocrinology and Nutrition of the European Society of Intensive Care Medicine. Crit Care. 2020 May 15;24(1):224. doi: 10.1186/s13054-020-02889-4. PMID 32414423